CLINICAL TRIAL: NCT06492239
Title: Emergency Stroke Unit for Acute Cerebrovascular Events--A Prospective, Multicenter, Week-wise Randomized, Controlled Trial ( ESU-ACE-A )
Brief Title: Emergency Stroke Unit for Acute Cerebrovascular Events ( ESU-ACE-A )
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yongjun Wang, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-131-02-A
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke, Acute
Keywords: Emergency stroke unit; Low-field magnetic resonance imaging; Reperfusion therapy; Intravenous thrombolysis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergency Stroke Unit based on 0.23-T MRI (Experimental): The participants with hyperacute ischemic stroke (symptoms onset ≤4.5 h) who are eligible to receive reperfusion therapy will be managed by Emergency Stroke Unit process based on low-field magnetic resonance imaging.
  Interventions: Combination Product: Emergency Stroke Unit based on 0.23-T MRI
- Standard stroke unit adherent to guidelines (Placebo Comparator): The participants with hyperacute ischemic stroke (symptoms onset ≤4.5 h) who are eligible to receive reperfusion therapy will be managed by standard stroke unit process adherent to guidelines.
  Interventions: Combination Product: Standard stroke unit adherent to guidelines

INTERVENTIONS:
Combination Product: Emergency Stroke Unit based on 0.23-T MRI — The participants with hyperacute ischemic stroke (symptoms onset ≤4.5 h) who are eligible to receive reperfusion therapy will be managed by Emergency Stroke Unit process based on low-field magnetic resonance imaging.
  Arms: Emergency Stroke Unit based on 0.23-T MRI
Combination Product: Standard stroke unit adherent to guidelines — The participants with hyperacute ischemic stroke (symptoms onset ≤4.5 h) who are eligible to receive reperfusion therapy will be managed by standard stroke unit process adherent to guidelines.
  Arms: Standard stroke unit adherent to guidelines

SUMMARY:
To compare the door-to-needle time of patients with hyperacute ischemic stroke (within 4.5 hours after the onset of symptoms) managed in a standard stroke unit adherent to guidelines versus managed in Emergency Stroke Unit (a new stroke unit based on low-field magnetic resonance imaging).

DETAILED DESCRIPTION:
Intravenous thrombolysis is an effective reperfusion therapy for patients with acute ischemic stroke. Faster door-to-needle time (DNT) is associated with significantly better clinical outcomes. With the development of low-field magnetic resonance imaging, it is poised to play an increasingly significant role in the early diagnosis and management of acute ischemic stroke. This prospective, multicenter, week-wise randomized controlled trial will compare the door-to-needle time of patients with hyperacute ischemic stroke (within 4.5 hours after the onset of symptoms) managed in a standard stroke unit adherent to guidelines versus managed in Emergency Stroke Unit (a new stroke unit based on low-field magnetic resonance imaging).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Can be treated within 4.5 hours of symptoms onset*(*Symptom onset is defined by the "last seen normal" principle);
3. Presenting with ischemic stroke symptoms;
4. Pre-stroke mRS score 0-1;
5. Baseline NIHSS score ≥ 5;
6. Eligible for rt-PA/TNK thrombolysis;
7. Informed consent signed.

Exclusion Criteria:

1. Baseline NIHSS score < 5;
2. Unable to undergo MRI because of claustrophobia;
3. Patients with cardiac pacemaker/brain pacemaker/insulin pump implantation;
4. Definite contraindication for rt-PA/TNK thrombolysis;
5. Patients with postictal hemiparesis (Todd's paralysis) or those with concomitant neurological/psychiatric conditions who are unable or unwilling to cooperate;
6. Pregnant women, nursing mothers, or reluctance to use effective contraceptive measures during the period of trial;
7. Participation in other interventional randomized clinical trials within 3 months before enrollment;
8. Patients deemed unsuitable for participation in this trial by the investigator or those for whom participation in this trial may result in greater risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Door-to-needle time | Door-to-needle time
  The time from emergency department arrival to the start of intravenous thrombolysis.

SECONDARY OUTCOMES:
The utility-weighted modified Rankin Scale (uw-mRS) at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).
  The utility-weighted modified Rankin Scale (uw-mRS) at 14±2 days (or at discharge, whichever occurs first). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Ordinal (shift) analysis of modified Rankin Scale (mRS) at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).
  Ordinal (shift) analysis of modified Rankin Scale (mRS) at 14±2 days (or at discharge, whichever occurs first). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Excellent functional outcome (Modified Rankin Scale score, mRS 0-1) at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).
  Excellent functional outcome (Modified Rankin Scale score, mRS 0-1) at 14±2 days (or at discharge, whichever occurs first). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Good functional outcome (Modified Rankin Scale score, mRS 0-2) at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).
  Good functional outcome (Modified Rankin Scale score, mRS 0-2) at 14±2 days (or at discharge, whichever occurs first). Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
The utility-weighted modified Rankin Scale (uw-mRS) at 90±7 days. | at 90±7 days.
  The utility-weighted modified Rankin Scale (uw-mRS) at 90±7 days. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Ordinal (shift) analysis of modified Rankin Scale (mRS) at 90±7 days. | at 90±7 days.
  Ordinal (shift) analysis of modified Rankin Scale (mRS) at 90±7 days. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Excellent functional outcome (Modified Rankin Scale score, mRS 0-1) at 90±7 days. | at 90±7 days.
  Excellent functional outcome (Modified Rankin Scale score, mRS 0-1) at 90±7 days. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
Good functional outcome (Modified Rankin Scale score, mRS 0-2) at 90±7 days | at 90±7 days.
  Good functional outcome (Modified Rankin Scale score, mRS 0-2) at 90±7 days. Scores on the modified Rankin scale range from 0 (no neurologic deficit) to 6 (death).
The time from symptoms onset to intravenous thrombolysis decision. | The time from symptoms onset to intravenous thrombolysis decision.
The time from emergency department arrival to intravenous thrombolysis decision. | The time from emergency department arrival to intravenous thrombolysis decision.
Symptomatic intracranial hemorrhages (according to the ECASS III criteria) within 36 hours. | within 36 hours.
  Symptomatic intracranial hemorrhages within 36 hours (sICH definition: according to the ECASS III criteria: any apparently extravascular blood in the brain or within the cranium that was associated with clinical deterioration, as defined by an increase of 4 points or more in the score on the NIHSS, or that led to death and that was identified as the predominant cause of the neurological deterioration).
Symptomatic intracranial hemorrhages (according to the ECASS III criteria) at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).
  Symptomatic intracranial hemorrhages at 14±2 days (or at discharge, whichever occurs first) (sICH definition: according to the ECASS III criteria: any apparently extravascular blood in the brain or within the cranium that was associated with clinical deterioration, as defined by an increase of 4 points or more in the score on the NIHSS, or that led to death and that was identified as the predominant cause of the neurological deterioration).
Mortality at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).
Adverse events at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).
Serious adverse events at 14±2 days (or at discharge, whichever occurs first). | at 14±2 days (or at discharge, whichever occurs first).

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No